CLINICAL TRIAL: NCT06206564
Title: A Phase II Double Blind, Placebo-controlled, Randomized Trial of Artesunate Ointment for the Treatment of HIV-negative Patients With Anal High-grade Squamous Intraepithelial Lesions (Anal HSIL)
Brief Title: Artesunate Ointment for the Treatment of Anal HSIL in HIV-negative Participants
Acronym: ART-AIN IIB-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Frantz Viral Therapeutics, LLC (Industry)
Collaborators: Laser Surgery Care, LLC (Unknown); Anal Dysplasia Clinic MidWest (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ART-AIN IIB-2
Record Dates: First submitted 2024-01-03; First posted 2024-01-16 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Anal High-grade Squamous Intraepithelial Lesion; Anal HSIL; Anal HPV Infection; AIN
Keywords: intra-anal; topical; non-surgical
MeSH Terms: interventions — artesunic acid; artenimol; artemisinin

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled randomized trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Artesunate (Experimental)
  Interventions: Drug: Artesunate ointment
- Placebo ointment (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Artesunate ointment — Four 5-day cycles of artesunate ointment given at weeks 0, 2, 4, 6
  Other Names: Artesunic acid; Dihydroartemisinin (DHA); Artemisinin
  Arms: Artesunate
Drug: Placebo — Four 5-day cycles of placebo ointment given at weeks 0, 2, 4, 6
  Other Names: placebo ointment
  Arms: Placebo ointment

SUMMARY:
This is a phase II double blind, placebo-controlled, randomized study of artesunate ointment for the treatment of HIV-negative men and women who have anal high grade squamous intraepithelial lesions (anal HSIL)

DETAILED DESCRIPTION:
Eligible participants in this study are randomized 2:1 to receive either artesunate or placebo ointment for the treatment of anal HSIL. Both groups receive four 5-day cycles of ointment, at weeks 0, 2, 4, and 6. Participants are followed closely with anoscopy or high resolution anoscopy (HRA) at weeks 8, 18, 30, and 42. After the week 18 HRA visit, participants who have at least partial response will be followed with HRA at week 30.

Participants who are found to be non-responders at week 18 will undergo standard of care ablation.

Participants who are found to have anal HSIL at weeks 30 or 42 will be followed according to standard of care procedures.

Primary Objective: To evaluate the complete and partial histopathologic response to four 5-day cycles of artesunate ointment in adult patients with biopsy-proven HPV-associated intra-anal HSIL (18 weeks).

Secondary Objectives:

Efficacy:

To evaluate the viral clearance after four 5-day cycles of artesunate ointment To evaluate complete and partial intra-anal response To evaluate complete and partial peri-anal response To evaluate persistence of response throughout the study window

Safety:

To evaluate the safety of artesunate ointment for the treatment of intra-anal HSIL.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women age ≥ 18 years
* Capable of informed consent
* Biopsy-confirmed intra-anal high-grade dysplasia (AIN 2, AIN 3, anal HSIL) by HRA.
* Positive anal human papillomavirus (HPV) test.
* Women of childbearing potential agree to use birth control for the duration of the study.
* Laboratory values at Screening of:

  1. Serum alanine transaminase (SGPT/ALT) < 5 x upper limit of normal (ULN)
  2. Serum aspartate transaminase (SGOT/AST) < 5 x ULN
  3. Serum Bilirubin (total) < 2.5 x ULN
  4. Serum Creatinine ≤ 1.5 x ULN
* Electrocardiogram (ECG) with no clinically significant findings as assessed by the Investigator.
* Weight ≥ 50kg

Exclusion Criteria:

* Pregnant and nursing women
* Diagnosis of low-grade anal dysplasia (AIN 1, LSIL), without the concomitant diagnosis of anal HSIL, by HRA
* Concurrent anal, vulvar, cervical, or penile cancer
* HIV-seropositivity
* Currently receiving systemic chemotherapy or radiation therapy for another cancer.
* Patients who are on medical treatment with systemic immunosuppressants or steroids (e.g., active autoimmune disease). Participants using nasal steroid treatments for allergic conditions may participate in the study.
* Concomitant use of strong UGT (Uridine-diphosphate-glucuronosyltransferase) inhibitors
* Concomitant use of imiquimod or 5-fluorouracil (5-FU) for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete and partial response by week 18 | 18 weeks
  Number of participants with complete and partial response after four 5-day cycles of artesunate ointment

SECONDARY OUTCOMES:
HPV clearance | 42 weeks
  Number of participants who do not have detectable HPV infection
Complete and partial response after week 18 | 30 weeks
  Number of participants with complete and partial response after week 18
Complete and partial peri-anal response after intra-anal ointment application | 42 weeks
  Number of participants who have complete and partial peri-anal response after 4 5-day cycles of intra-anal ointment
Persistence of response | 42 weeks
  Number of participants who have complete response and do not have recurrence of anal HSIL

OTHER OUTCOMES:
Safety of intra-anal artesunate ointment | 42 weeks
  Number of participants who do not have any drug-related serious adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Anal Dysplasia Clinic MidWest, Chicago, Illinois
  - Laser Surgery Care, New York, New York

IPD SHARING:
Plan to Share IPD: No
No protected health information (PHI) will be shared with other researchers.